CLINICAL TRIAL: NCT05559177
Title: An Open, Dose-escalation Clinical Study of Chimeric Exosomal Tumor Vaccines for Recurrent or Metastatic Bladder Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDZJ-01
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Recurrent or Metastatic Bladder Cancer
MeSH Terms: conditions — Recurrence; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of recurrent or metastatic bladder cancer (Experimental): Lack of conventional effective treatment, failure or recurrence of treatment with conventional methods (surgery, chemotherapy, radiotherapy, immune checkpoint inhibitors, targeted therapy, etc.), or refusal of conventional treatment
  Interventions: Biological: Chimeric exosomal tumor vaccines

INTERVENTIONS:
Biological: Chimeric exosomal tumor vaccines — Tumor cells (lesion site) were isolated from bladder cancer patients, and bladder cancer nuclei were extracted. Monocytes were isolated from peripheral blood of this patient and induced in vitro to obtain APC (DC or macrophage). Apc-tumor chimeric cells were constructed and stimulated with immune stimulator. Chimeric exosomal vaccines were extracted from cell supernatants by differential and hypervelocity centrifugation

SUMMARY:
1. Based on the applicant's previous work and combined with the clinical medical resources of our unit, tumor cells were isolated from the lesion site of cancer patients, dendritic cells or macrophages were isolated from peripheral blood, and personalized chimeric exosome vaccine was prepared for patients.
2. To evaluate the safety and tolerability of multiple administration of chimeric exosome vaccine in subjects with hatching or metastatic bladder cancer, explore the maximum tolerated dose (MDT) and dose-limiting toxicity (DLT) in humans, and recommend the safe dose range for the subsequent extended trials and subsequent clinical studies of this product.
3. To reveal the "double-effect" improvement mechanism of chimeric exosome vaccine on the activation of immune response and the microenvironment of bladder cancer lesions, improve the anti-recurrence treatment effect of bladder cancer, and realize the clinical transformation of "double-target and double-effect" chimeric exosome vaccine in the field of individualized precision treatment of bladder cancer patients.
4. To explore the clinical application value of this tumor therapeutic vaccine by using the T-cell receptor immunoomics and immunomolecular evaluation technology platform established by previous researchers, and to provide preliminary clinical research results for further vaccine development.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bladder cancer confirmed by histopathology and/or cytology;
2. Age ≥18 years old and ≤85 years old, both sexes;
3. ECOG score of general physical condition 0 ~ 2 points;
4. The expected survival time is at least 3 months.
5. Lack of conventional effective treatment, failure or recurrence after conventional treatment (surgery, chemotherapy, radiotherapy, immune checkpoint inhibitors, targeted therapy, etc.), or refusal of conventional treatment;
6. According to RECIST criteria, at least one measurable objective tumor index (target lesion ≥10mm detected by spiral CT);
7. At baseline, WBC≥3.5×109/L, Hb≥90g/L, PLT≥80×109/L;
8. Subjects must have adequate organ function and the following laboratory tests during the screening period must be met:

   A) Absolute neutrophil count (ANC)≥1.5×109 /L, platelet (PLT)≥ 80×109 /L, hemoglobin (Hb)≥ 85g/L;

   B) Serum creatinine (Cr) and blood urea nitrogen (BUN) within 1.5 times the upper limit of normal values;

   C) Serum total bilirubin (TBIL) ≤ 2 times of the upper limit of normal;

   D) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times of the upper limit of normal values; Subjects with liver metastases were no more than 5 times the upper limit of normal;

   E) Activated partial thromboplastin time (APTT) and prothrombin time (PT) were within 1.5 times of the upper limit of normal values;
9. Eligible fertile patients (male and female) must consent to use a reliable contraceptive method (hormonal or barrier or abstinence) with their partner during the trial and for at least 180 days after the last dose; Women of childbearing age must have a negative urinary pregnancy test within 7 days before enrollment;
10. Subject signed informed consent voluntarily and expected compliance was good.

Exclusion Criteria:

1. Severe infection and other serious complications;
2. The patient has a previous or current primary malignancy associated with other sites, excluding effectively treated non-malignant melanoma skin cancer, carcinoma in situ of the cervix, or other malignancy that has been potentially curable with effective treatment and has been in remission for at least 5 years;
3. Patients with a history of autoimmune diseases, including but not limited to multiple sclerosis, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, but not vitiligo;
4. Patients with systemic corticosteroid or other immunosuppressive hormone therapy can be treated with prednisone < 0.5 mg/kg/day (maximum cell number group 40 mg/day) or other similar drugs in the equivalent cell number group, inhaled corticosteroid hormones can be used for chronic obstructive pulmonary disease (COPD) or topical use
5. Patients who have undergone major organ transplants;
6. Patients with active bleeding or severe coagulopathy;
7. Patients with active pulmonary tuberculosis and strong positive OT test;
8. Patients with previous severe interstitial lung changes (as determined by the investigator);
9. Subjects with any severe and/or uncontrolled disease, including:

   A) poor control of hyperbole (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥100mmHg);

   B) Patients with grade I or higher myocardial ischemia or infarction, arrhythmias (including QTc≥ 450ms in men and QTc≥470ms in women), and congestive heart failure grade ≥2 (NYHA classification);

   C) Active or uncontrolled severe infection (≥CTCAE grade 2 infection);

   D) Patients with previous organ transplantation, bone marrow transplantation (hematopoietic stem cell transplantation) and severe immune deficiency;

   E) Urine routine indicated urinary protein ≥++, and confirmed 24-hour urinary protein quantification > 1.0 g;
10. Four weeks before the first drug administration, antitumor therapy was performed, including endocrine, chemotherapy, radiotherapy, targeted therapy, immunotherapy and antitumor Chinese medicine therapy; For subjects receiving nitrolurea and mitomycin chemotherapy, discontinuation was within 6 weeks;
11. Had received a prophylactic or attenuated or therapeutic vaccine within 4 weeks before the first dose;
12. Toxicity after previous antitumor therapy has not recovered to CTCAE 5.0 grade 0 or level 1;
13. Current active hepatitis B, active hepatitis C, immunodeficiency virus, or other active infection of clinical significance;
14. Patients who had undergone tertiary surgery or unhealed surgical wounds 4 weeks before enrollment;
15. Participated in other clinical trials within four weeks before enrollment;
16. Pregnant or lactating women and those who plan to give birth within six months (male or female);
17. In the judgment of the investigator, the subject is not suitable to participate in the trial for any reason -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | 24 months
  The percentage of patients with CR and PR in the total number of patients in the same period
Overall survival(OS) | 24 months
  From the starting date of the enrollment until the date of the first documented disease progression or the date of the death from any cause,whichever comes first
Safty(adverse events) | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Pudong Medical Center, Shanghai, China